CLINICAL TRIAL: NCT05179993
Title: Detection of Microplastics in Human Granulosa Cells and in the Follicular Fluid of Women Undergoing Intracytoplasmic Sperm Injection (ICSI) Treatment
Brief Title: Detection of Microplastics in Human Granulosa Cells and in the Follicular Fluid of Women Undergoing ICSI Treatment
Acronym: MP2021
Status: Recruiting | Type: Observational
Sponsor: Infertility Treatment Center Dortmund (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: Microplastic
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Female Infertility; Environmental Exposure
Keywords: Microplastics; Follicular Fluid; Granulosa Cells
MeSH Terms: conditions — Infertility, Female | interventions — Microplastics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human granulosa cells and human follicular fluid of women undergoing ICSI Treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: Proof of principle Study group: detection of microplastics in human granulosa cells and in the follicular fluid of women undergoing intracytoplasmic sperm injection (ICSI) treatment
  Interventions: Other: Microplastics

INTERVENTIONS:
Other: Microplastics — Detection of microplastics as a yes/no value

SUMMARY:
Plastic products have been used ubiquitously in the modern world for many decades - for example as packaging materials, textile fibers or molded parts. The general use and especially the improper disposal lead to enormous environmental pollution almost everywhere on earth.

Microplastics mainly originate from fragmentation of larger plastic objects or can be produced directly for the use in e.g. cosmetics or industrial dyes.

Microplastics have already been detected in fresh- and seawater, soil, food, but also in human blood and urine. The accumulation of microplastics in ovarian and testicular tissue in humans has not yet been investigated.

DETAILED DESCRIPTION:
Plastic products have been used ubiquitously in the modern world for many decades - for example as packaging materials, textile fibers or molded parts. The general use and especially the improper disposal lead to enormous environmental pollution almost everywhere on earth. In particular microplastics, by definition plastic particles with a diameter of less than 5mm, could pose a hazard to animals, humans and nature. Microplastics mainly originate from fragmentation of larger plastic objects or can be produced directly for the use in e.g. cosmetics or industrial dyes.

Microplastics have already been detected in fresh- and seawater, soil, food, but also in human blood and urine. The accumulation of microplastics in ovarian and testicular tissue in humans has not yet been investigated.

The presence of microplastics in reproductive tissue could also have negative consequences for reproduction. In oysters, waterfleas and mice, an impairment of reproduction due to the bioaccumulation of microplastics has already been described. Overall, current understanding of the effects of microplastics on human fertility and overall mammalian health is very limited.

Samples will be analyzed using Raman spectroscopy and scanning electron microscopy.

ELIGIBILITY:
Inclusion Criteria:

* The patients to be included should be ≥18 years of age undergoing an intracytoplasmic sperm injection (ICSI) treatment. There is no upper limit for patient age.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population is made up of patients from the Fertility Center Dortmund who have given their consent to the study after being informed by the attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of microplastics in human granulosa cells and in the Follicular fluid | 1 day (directly after oocyte pick-up)
  Detection of microplastics in human granulosa cells and in the Follicular fluid of women undergoing intracytoplasmic sperm injection (ICSI) treatment as a binary value (yes / no).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Dieterle, MD, Principal Investigator — Infertility Treatment Center Dortmund
Locations (1):
- Infertility treatment center Dortmund, Dortmund, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No